CLINICAL TRIAL: NCT06717022
Title: A Clinical Study of CHT102, a Universal Chimeric Antigen Receptor T-Cell Immunotherapy(U CAR-T) for Mesothelin(MSLN) Positive Advanced Solid Tumors: a Single-arm, Open-label, Dose Escalation and Expansion Clinical Study
Brief Title: A Clinical Study of CHT102 in Mesothelin Positive Advanced Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Nanjing Calmhome Cell and Gene Engineering Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHT102SIIT-01
Record Dates: First submitted 2024-11-21; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Mesothelin Positive Tumors
Keywords: CHT102, a U CAR-T therapy for MSLN-positive advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHT102 allogeneic CAR T cells (Experimental): In the dose escalation phase of this study, one alternative dose and 4 dose groups (calculated by the number of CAR-positive T cells) were planned, each treatment lasted 28 days, and UCAR-T cells were transfused three times, respectively on D1, D5, and D9. The single dose within the group was fixed, and the dose between the groups was escalating dose. Each infusion dose was 2.5×106/kg (optional), 5×106/kg, 1×107/kg, 2×107/kg, and 3×107/kg, with a dose error of 20% allowed.
  Interventions: Biological: CHT102 allogeneic CAR T cells

INTERVENTIONS:
Biological: CHT102 allogeneic CAR T cells — CHT102 allogeneic CAR T cells

SUMMARY:
Objectives of Study：In this study investigators plan to evaluate the safety and efficacy of MSLN-targeting Universal Chimeric Antigen Receptor T-Cell Immunotherapy(U CAR-T) in the treatment of MSLN-positive advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent document；
* Age ≥18 years old, male or female；
* Histopathological confirmed advanced or metastatic solid tumors failed to at least standard first-line therapy or initially diagnosed advanced solid tumors that have no National Comprehensive Cancer Network (NCCN ）guideline recommended standard first-line therapy；
* Histopathology or cytology (paraffin section or fresh biopsy tumor tissue specimen) diagnosed as advanced/metastatic solid tumor (positive tumor MSLN expression (tumor MSLN positive (IHC 2+) confirmed by histology or pathology));
* At least one measurable lesion at baseline per RECIST version 1.1；
* The expected survival time is more than 12 weeks;
* ECOG(American Eastern Oncology Consortium) 0-1 points;
* The function of important organs is basically normal;
* The investigator determines that the patient must have fully recovered from previous treatment toxicity to ≤ grade 1, except in the following cases: a. Hair loss; b. Pigmentation; c. Long-term toxicity caused by radiotherapy, which could not be recovered according to the investigators; d. Platinum induced grade 2 or lower neurotoxicity (CTCAE 5.0);
* Subjects agree to use reliable and effective contraceptive methods for contraception within
* 6 months after signing the informed consent form to receiving CAR-T cell infusion (excluding rhythm contraception).

Exclusion Criteria:

* Received any experimental drug treatment or used experimental devices within 28 days;
* Received anti-tumor therapy such as chemotherapy and targeted therapy within 4 weeks;
* Received cell therapy products other than MSLN targets within 1 month;
* Patients who have previously received other cell therapy products should be tested for RCL(Replication Competent Retrovirus ) during the screening period if any test result is positive;
* Received chemotherapy other than lymphocyte clearance chemotherapy within 14 days prior to CHT102 infusion;
* Received systemic corticosteroid therapy at doses greater than 10 mg/day prednisone (or equivalent doses of other corticosteroids) within 2 weeks；
* Patients receiving oral or intravenous anticoagulant therapy within 7 days prior to CHT102 cell infusion;
* Prior organ allograft transplantations or allogeneic hematopoietic stem cell transplantation;
* Patients with immune deficiency or autoimmune diseases, or who require immunosuppressants;
* Vaccination within 14 days of study enrollment, or who required live vaccine immunization during the study period;
* Active/symptomatic central nervous system metastases or meningeal metastases at the time of screening; subjects with brain metastases who have been treated must be confirmed to have no imaging evidence of progression ≥ 4 weeks after the end of treatment before they can be enrolled;
* Serious or uncontrollable systemic disease or any unstable systemic disease, including but not limited to uncontrolled hypertension, uncontrolled hyperglycemia, liver and kidney insufficiency or metabolic disease, central nervous system disease, etc;
* Have any of the following heart conditions:
* New York Heart Association (NYHA) stage III or IV congestive heart failure;
* Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months before enrollment;
* Clinically significant ventricular arrhythmia,
* echocardiography showed cardiac ejection fraction<50%, QTc (male)>450 ms，QTc (female)>470 ms；;
* Pregnant, lactating, or breastfeeding females;
* Patients with poor control of thoracoabdominal water;
* Other investigators deem it inappropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2039-05 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLTs) occurence | Baseline up to 28 days after U CAR-T infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Objective Response Rate | At 4 weeks, and overall
  The total response rate after 90 days of treatment with study drug.
Progression-free survival | Assessed up to 6 months
  Progression-free survival rate following drug therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China